CLINICAL TRIAL: NCT04318444
Title: Hydroxychloroquine Post Exposure Prophylaxis (PEP) for Household Contacts of COVID-19 Patients: A NYC Community-Based Randomized Clinical Trial
Brief Title: Hydroxychloroquine Post Exposure Prophylaxis for Coronavirus Disease (COVID-19)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The Institutional Review Board closed the study
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAS9676
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; Corona Virus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxychloroquine (Experimental): Two tablets (400mg) twice daily on day 1; for days 2-5, they will be instructed to take one tablet (200mg) twice daily.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Two tablets (400mg) twice daily on day 1; for days 2-5, they will be instructed to take one tablet (200mg) twice daily.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — Two tablets (400mg) twice daily on day 1; for days 2-5, they will be instructed to take one tablet (200mg) twice daily.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo oral tablet — Two tablets (400mg) twice daily on day 1; for days 2-5, they will be instructed to take one tablet (200mg) twice daily.
  Other Names: Placebo Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that post-exposure prophylaxis with hydroxychloroquine will reduce the symptomatic secondary attack rate among household contacts of known or suspected COVID-19 patients.

DETAILED DESCRIPTION:
COVID-19 is a massive threat to public health worldwide. Current estimates suggest that the novel coronavirus (SARS-CoV-2) is both highly contagious (estimated reproductive rate, 2-3) and five to fifty-fold more lethal than seasonal influenza (estimated mortality rate, 0.5-5%). Interventions to decrease the incidence and severity of COVID-19 are emergently needed.

Hydroxychloroquine (brand name, Plaquenil), an inexpensive anti-malarial medication with immunomodulatory effects, is a promising therapy for COVID-19. Chloroquine, a related compound with a less favorable toxicity profile, has shown benefit in clinical studies conducted in approximately one-hundred SARS-CoV-2 infected patients. In vitro, hydroxychloroquine has been recently shown to have greater efficacy against SARS-CoV-2 versus chloroquine.

Currently, there is no established post-exposure prophylaxis for persons at high risk of developing COVID-19. Hydroxychloroquine (brand name, Plaquenil), is a medicine that has been found to be effective against the novel coronavirus in some recent experiments. Previously, hydroxychloroquine has been safety used to prevent malaria or to treat autoimmune diseases.

This study will test if hydroxychloroquine may be used to prevent the development of COVID-19 symptoms in persons who live with an individual who has been diagnosed with COVID-19. If hydroxychloroquine is shown to reduce the risk of developing symptoms of COVID-19 among people at high risk of infection, this could help to reduce the morbidity and mortality of the COVID-19 epidemic.

This is a trial of hydroxychloroquine PEP among adult household contacts of COVID-19 patients in New York City (NYC). The trial will be initiated at NewYork-Presbyterian (NYP)/Columbia University Irving Medical Center (CUIMC).

ELIGIBILITY:
Inclusion Criteria:

* Household contact of index case: currently residing in the same household as an individual evaluated at NYP via outpatient, emergency department (ED), or inpatient services who (1) test positive for COVID-19, or (2) are defined as suspected cases, or persons under investigations (PUI), by the treating physician.
* Willing to take study drug as directed for 5 days.

Exclusion Criteria:

* Age <18 years old
* Suspected or confirmed current COVID-19, defined as: (1) temperature > 38 Celsius; (2) cough; (3) shortness of breath; (4) sore throat; or, if available (not required), (5) positive confirmatory testing for COVID-19
* Suspected or confirmed convalescent COVID-19, defined as any of the above symptoms within the prior 4 weeks.
* Inability to take medications orally
* Inability to provide written consent
* Known sensitivity/allergy to hydroxychloroquine
* Current use of hydroxychloroquine for another indication
* Pregnancy
* Prior diagnosis of retinopathy
* Prior diagnosis of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Major comorbidities increasing risk of study drug including: i. Hematologic malignancy, ii. Advanced (stage 4-5) chronic kidney disease or dialysis therapy, iii. Known history of ventricular arrhythmias, iv. Current use of drugs that prolong the QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-29 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon T. Giles, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akhtar S, Das JK, Ismail T, Wahid M, Saeed W, Bhutta ZA. Nutritional perspectives for the prevention and mitigation of COVID-19. Nutr Rev. 2021 Feb 11;79(3):289-300. doi: 10.1093/nutrit/nuaa063. PMID 33570583

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 8 completers out of 10 enrolled/consented. 2 participants withdrew consent prior to initiating study intervention.
Groups:
- Hydroxychloroquine Group: Participants will take 2 tablets (400mg) of hydroxychloroquine orally twice daily on day 1; for days 2-5, they will be instructed to take 1 tablet (200mg) twice daily.
- Placebo Group: Participants will take 2 tablets (400mg) of placebo orally twice daily on day 1; for days 2-5, they will be instructed to take 1 tablet (200mg) twice daily.
Period: Overall Study
Arm/Group | Hydroxychloroquine Group | Placebo Group
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 out of 10 consented participants withdrew consent prior to initiating study intervention.
  Due to the low number of participants per group, baseline characteristics are presented as one arm to protect the confidentiality of the participants.
Groups:
- Hydroxychloroquine/Placebo Group: Participants will take 2 tablets (400mg) of either hydroxychloroquine or placebo orally twice daily on day 1. For days 2-5, they will be instructed to take 1 tablet (200mg) of either hydroxychloroquine or placebo orally twice daily.
Arm/Group | Hydroxychloroquine/Placebo Group
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic, Lab-confirmed COVID-19.
Description: This is defined as either 1. COVID-19 infection confirmed within 14 days of enrollment, following self-report of COVID-19 symptoms to the research study; OR, 2. COVID-19 infection confirmed within 14 days of enrollment, with self-report of COVID-19 symptoms to a treating physician.
Time Frame: Date of enrollment to 14 days post-enrollment date
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine Group | Placebo Group
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days
Arm/Group | Hydroxychloroquine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT04318444/Prot_SAP_000.pdf